CLINICAL TRIAL: NCT06497231
Title: Clinical and Periodontal Evaluation of Deep Marginal Elevation for Proximal Carious Lesions Restored with Bioactive Giomer Versus Nanohybrid Resin Composite: Two Years Randomized Trial
Brief Title: Evaluation of Bioactive Giomer Material Versus Nanohybrid Resin Composite in Deep Marginal Elevation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Samir Ashraf Fayez Rostom, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Giomer in DME
Record Dates: First submitted 2024-07-04; First posted 2024-07-11 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-06

CONDITIONS: Deep Caries; Dental Caries
Keywords: Deep marginal elevation; Giomer
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Bioactive Giomer Material (Active Comparator): Deep margin elevation and subsequent restoration will be done using bioactive giomer material
  Interventions: Other: Beautifil II LS
- Nanohybrid resin composite (Active Comparator): Deep margin elevation and subsequent restoration will be done using nanohybrid resin composite
  Interventions: Other: Nanohybrid resin composite material

INTERVENTIONS:
Other: Beautifil II LS — Beautifil II LS is a low shrinkage bioactive giomer resin composite.
  Arms: Bioactive Giomer Material
Other: Nanohybrid resin composite material — Nanohybrid resin composite is a type of restorative material that features nano-sized fillers as a main component.
  Arms: Nanohybrid resin composite

SUMMARY:
This study will be conducted to evaluate the clinical, radiographic and periodontal performance of bioactive Giomer compared to nanohybrid resin composite restoration in deep subgingival proximal cavities extending below the CEJ over a period of 24 months.

DETAILED DESCRIPTION:
Background and rationale:

Recent development in different adhesive techniques and materials has led clinicians to attempt restoring teeth with subgingival defects below the cemento-enamel junction (CEJ). Deep marginal elevation (DME) or cervical margin relocation (CMR) is a procedure that involves raising the proximal margin of the tooth defect with direct composite to promote isolation and restoration using direct, semi-direct or indirect techniques. A high level of knowledge and clinical expertise are necessary to perform such procedure in a predictable way in addition to meticulous attention to the supracrestal tissue attachment or the biological width which consists of junctional epithelium and supracrestal connective tissue attachment.

Research question:

In young and middle-aged patients having deep subgingival proximal cavities extending below CEJ, will the bioactive Giomer show similar clinical, radiographic and periodontal performance compared to nanohybrid resin composite over 2 years follow up?

Statement of the problem:

Carious lesions that extend in subgingival areas present several difficulties for the clinician. Firstly, applying rubber dam in deep cavities and the process of trying to obtain a gingival margin free of caries are very challenging. Secondly, there is a great biological concern to master the subgingival restoration reaction with the adjacent periodontal tissues. Obtaining a healthy periodontal status after treatment has long been a challenging endeavor in the restorative dentistry. Lastly, bonding to deep, carious, and moist dentin surrounded by cementum is inherently suboptimal. To overcome these problems, many techniques and materials were presented to deal with such complex restorative situations. Because of their chemical adherence to the tooth structure, fluoride release and hydrophilicity glass ionomer cements are a reliable option for cementum margins and deep dentin bonding. Marginal defects appearing at the cervical margins due to the solubility property of the material was the main problem the dentist faced in these situations. On the other hand, resin composites are a dependable choice in these circumstances due to their higher mechanical qualities and the way their composition has improved, however, poor material bonding in subgingival margins along with high polymerization stresses associated with them have made it a very complicated procedure.

Rationale for conducting the research:

The use of fluoride releasing dental materials in deep carious lesions was explored before to remineralize the surrounding tooth structure and allow for a more durable restoration with increased resistance to the development of secondary caries. The introduction of Giomers, which combines resin composite and glass ionomer modes of action by Shofu, (Inc.) in the early 2000s was due to the revolutionary surface prereacted glass-ionomer (S-PRG) filler technology that allowed for improved resistance to recurrent caries development. Therefore, this type of bioactive system, adhesive and restoring materials, was claimed to enhance the outcome of deep subgingival restoration clinically, periodontally, and radiographically.

ELIGIBILITY:
Inclusion Criteria:

1. Young and middle aged patients (20-50)
2. Good or moderate oral hygiene (plaque index 0 or 1 )
3. Patient approval
4. Absence of parafunctional habits and/or bruxism

Exclusion Criteria:

1. Patients with known allergic or adverse reaction to the tested materials.
2. Systematic disease that may affect participation.
3. Xerostomic patients.
4. Patients with active periodontal disease.
5. Heavy smokers

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Post-operative sensitivity | Baseline (1 week after intervention), 6 months, 12 months and 24 months
  Restorations will be assessed by testing of irritability of the pulpal nerve on cold, e.g., with dry ice or cold spray, in comparison to the reaction of a contralateral, sound, and unrestored tooth.

SECONDARY OUTCOMES:
Marginal adaptation | Baseline (1 week after intervention), 6 months, 12 months and 24 months
  Method of restorations assessment will be Tactile using different sized explorers. Assessment will be done using FDI criteria and recorded as scores from 1 to 5, where scores from 1 to 5 will indicate clinically excellent/very good, clinically good, clinically satisfactory, clinically unsatisfactory and clinically poor respectively.
Occurrence of caries | Baseline (1 week after intervention), 6 months, 12 months and 24 months
  Method of restorations assessment will be Tactile using different sized explorers. Assessment will be done using FDI criteria and recorded as scores from 1 to 5, where scores from 1 to 5 will indicate clinically excellent/very good, clinically good, clinically satisfactory, clinically unsatisfactory and clinically poor respectively.
Proximal Contact | Baseline (1 week after intervention), 6 months, 12 months and 24 months
  Method of restorations assessment will be tactile using unwaxed dental floss to evaluate proximal contact tightness. Assessment will be done using FDI criteria and recorded as scores from 1 to 5, where scores from 1 to 5 will indicate clinically excellent/very good, clinically good, clinically satisfactory, clinically unsatisfactory and clinically poor respectively.
Plaque Index | Baseline (1 week after intervention), 6 months, 12 months and 24 months
  The Plaque Index (PI) is a clinical tool used by dentists to assess the presence and severity of dental plaque accumulation on the teeth. It is scored on a scale of 0 to 3:
  0: No plaque present.
  1. A thin film of plaque visible only with a probe or at the gingival margin.
  2. Moderate plaque accumulation visible to the naked eye.
  3. Heavy plaque accumulation visible on the tooth surface.
Gingival Index | Baseline (1 week after intervention), 6 months, 12 months and 24 months
  The Gingival Index (GI) is a clinical tool used to assess the health of the gums by evaluating the presence and severity of gingival inflammation.
  Gingival Index Scoring (0 to 3):
  The Gingival Index evaluates the gingiva (gums) at four sites per tooth (mesial, distal, buccal, and lingual). Each site is scored on a scale from 0 to 3:
  0: Normal gingiva - No inflammation, healthy gums.
  1. Mild inflammation - Slight redness, no bleeding on probing, no swelling.
  2. Moderate inflammation - Redness, slight swelling, and bleeding on probing.
  3. Severe inflammation - Redness, swelling, and bleeding even without probing; possibly ulcerated or visibly infected gums.
Interdental Pressure Index | Baseline (1 week after intervention), 6 months, 12 months and 24 months
  Apical pressure of a horizontally placed periodontal probe is applied to evaluate periodontal tissue response. It is negative when gingival tissues are firm, bleeding-free, and slightly ischemic by the stimulation; otherwise it is positive.
  It follows a negative or positive binary score.
Papillary bleeding on probing Index | Baseline (1 week after intervention), 6 months, 12 months and 24 months
  The Papillary Bleeding on Probing (PBI) Index is a clinical tool used to assess the presence of bleeding from the papillary gingiva (the area of gum tissue between the teeth) when a periodontal probe is gently inserted. This index helps evaluate the level of gingival inflammation and is commonly used in diagnosing gingivitis or early stages of periodontal disease.
  Scoring System: The PBI uses a simple scale to score bleeding, often as follows:
  0: No bleeding on probing - Healthy gingiva with no signs of inflammation.
  1. Bleeding on probing - A slight amount of bleeding from the papillary gingiva occurs within 15 seconds after probing.
  2. Bleeding on probing with immediate response - Bleeding is visible immediately after probing, indicating more significant inflammation.
  3. Spontaneous bleeding - Bleeding occurs without probing, indicating advanced gingival inflammation or active gum disease.
Probing Depth | Baseline (1 week after intervention), 6 months, 12 months and 24 months
Radiographic examination | Baseline (1 week after intervention), 6 months, 12 months and 24 months

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alleman DS, Magne P. A systematic approach to deep caries removal end points: the peripheral seal concept in adhesive dentistry. Quintessence Int. 2012 Mar;43(3):197-208. PMID 22299120
- [Background] Angerame D, De Biasi M. Do Nanofilled/Nanohybrid Composites Allow for Better Clinical Performance of Direct Restorations Than Traditional Microhybrid Composites? A Systematic Review. Oper Dent. 2018 Jul/Aug;43(4):E191-E209. doi: 10.2341/17-212-L. Epub 2018 Mar 23. PMID 29570022
- [Background] Bertoldi C, Monari E, Cortellini P, Generali L, Lucchi A, Spinato S, Zaffe D. Clinical and histological reaction of periodontal tissues to subgingival resin composite restorations. Clin Oral Investig. 2020 Feb;24(2):1001-1011. doi: 10.1007/s00784-019-02998-7. Epub 2019 Jul 8. PMID 31286261
- [Background] Blatz MB, Eggmann F. Deep Margin Elevation: Next-Level Adhesive Dentistry to Avoid Surgical Crown Lengthening. Compend Contin Educ Dent. 2023 Oct;44(9):530-531. PMID 37850958
- [Background] Bresser RA, Gerdolle D, van den Heijkant IA, Sluiter-Pouwels LMA, Cune MS, Gresnigt MMM. Up to 12 years clinical evaluation of 197 partial indirect restorations with deep margin elevation in the posterior region. J Dent. 2019 Dec;91:103227. doi: 10.1016/j.jdent.2019.103227. Epub 2019 Nov 4. PMID 31697971
- [Background] Checchi L, Montevecchi M, Marucci G, Checchi V. A proposed new index for clinical evaluation of interproximal soft tissues: the interdental pressure index. Int J Dent. 2014;2014:345075. doi: 10.1155/2014/345075. Epub 2014 Apr 1. PMID 24799903
- [Background] Cushley S, Duncan HF, Lappin MJ, Chua P, Elamin AD, Clarke M, El-Karim IA. Efficacy of direct pulp capping for management of cariously exposed pulps in permanent teeth: a systematic review and meta-analysis. Int Endod J. 2021 Apr;54(4):556-571. doi: 10.1111/iej.13449. Epub 2020 Dec 28. PMID 33222178
- [Background] Donly KJ, Segura A, Wefel JS, Hogan MM. Evaluating the effects of fluoride-releasing dental materials on adjacent interproximal caries. J Am Dent Assoc. 1999 Jun;130(6):817-25. doi: 10.14219/jada.archive.1999.0305. PMID 10377639
- [Background] Eggmann F, Ayub JM, Conejo J, Blatz MB. Deep margin elevation-Present status and future directions. J Esthet Restor Dent. 2023 Jan;35(1):26-47. doi: 10.1111/jerd.13008. Epub 2023 Jan 5. PMID 36602272
- [Background] El-Ma'aita AM, Radwan H, Al-Rabab'ah MA. Deep Margin Elevation - A Retrospective Clinical Study. J Adhes Dent. 2024 Apr 11;26:117-124. doi: 10.3290/j.jad.b5199089. PMID 38602235
- [Background] Ferrari M, Koken S, Grandini S, Ferrari Cagidiaco E, Joda T, Discepoli N. Influence of cervical margin relocation (CMR) on periodontal health: 12-month results of a controlled trial. J Dent. 2018 Feb;69:70-76. doi: 10.1016/j.jdent.2017.10.008. Epub 2017 Oct 20. PMID 29061380
- [Background] Gordan VV, Blaser PK, Watson RE, Mjor IA, McEdward DL, Sensi LG, Riley JL 3rd. A clinical evaluation of a giomer restorative system containing surface prereacted glass ionomer filler: results from a 13-year recall examination. J Am Dent Assoc. 2014 Oct;145(10):1036-43. doi: 10.14219/jada.2014.57. PMID 25270702
- [Background] Hickel R, Mesinger S, Opdam N, Loomans B, Frankenberger R, Cadenaro M, Burgess J, Peschke A, Heintze SD, Kuhnisch J. Correction to: Revised FDI criteria for evaluating direct and indirect dental restorations-recommendations for its clinical use, interpretation, and reporting. Clin Oral Investig. 2023 Jun;27(6):2593. doi: 10.1007/s00784-022-04851-w. No abstract available. PMID 36607493
- [Background] Ismail HS, Ali AI, El Mehesen R, Garcia-Godoy F, Mahmoud SH. Clinical evaluation of subgingival open sandwich restorations: 3-year results of a randomized double-blind trial. J Esthet Restor Dent. 2024 Apr;36(4):573-587. doi: 10.1111/jerd.13158. Epub 2023 Oct 30. PMID 37902283
- [Background] LOE H, SILNESS J. PERIODONTAL DISEASE IN PREGNANCY. I. PREVALENCE AND SEVERITY. Acta Odontol Scand. 1963 Dec;21:533-51. doi: 10.3109/00016356309011240. No abstract available. PMID 14121956
- [Background] Magne P. M-i-M for DME: matrix-in-a-matrix technique for deep margin elevation. J Prosthet Dent. 2023 Oct;130(4):434-438. doi: 10.1016/j.prosdent.2021.11.021. Epub 2021 Dec 25. PMID 34961611
- [Background] Deep Margin Elevation: A Paradigm Shift. American Journal of Esthetic Dentistry, 2, 86-96.
- [Background] Maran BM, de Geus JL, Gutierrez MF, Heintze S, Tardem C, Barceleiro MO, Reis A, Loguercio AD. Nanofilled/nanohybrid and hybrid resin-based composite in patients with direct restorations in posterior teeth: A systematic review and meta-analysis. J Dent. 2020 Aug;99:103407. doi: 10.1016/j.jdent.2020.103407. Epub 2020 Jun 9. PMID 32526348
- [Background] Muhlemann HR. Psychological and chemical mediators of gingival health. J Prev Dent. 1977 Jul-Aug;4(4):6-17. No abstract available. PMID 275483
- [Background] Bonding to caries-affected dentin. Japanese Dental Science Review, 47, 102-114.
- [Background] Neto CCL, das Neves AM, Arantes DC, Sa TCM, Yamauti M, de Magalhaes CS, Abreu LG, Moreira AN. Evaluation of the clinical performance of GIOMERs and comparison with other conventional restorative materials in permanent teeth: a systematic review and meta-analysis. Evid Based Dent. 2022 Aug 1. doi: 10.1038/s41432-022-0281-8. Online ahead of print. PMID 35915167
- [Background] Opdam NJM, VanBeek V, VanBeek W, Loomans BAC, Pereira-Cenci T, Cenci MS, Laske M. Long term clinical performance of 'open sandwich' and 'total-etch' Class II composite resin restorations showing proximal deterioration of glass-ionomer cement. Dent Mater. 2023 Sep;39(9):800-806. doi: 10.1016/j.dental.2023.07.001. Epub 2023 Jul 17. PMID 37468394
- [Background] Ozer F, Irmak O, Yakymiv O, Mohammed A, Pande R, Saleh N, Blatz M. Three-year Clinical Performance of Two Giomer Restorative Materials in Restorations. Oper Dent. 2021 Jan 1;46(1):E60-E67. doi: 10.2341/17-353-C. PMID 33882138
- [Background] Ramfjord SP. The Periodontal Disease Index (PDI). J Periodontol. 1967 Nov-Dec;38(6):Suppl:602-10. doi: 10.1902/jop.1967.38.6.602. No abstract available. PMID 5237683
- [Background] SILNESS J, LOE H. PERIODONTAL DISEASE IN PREGNANCY. II. CORRELATION BETWEEN ORAL HYGIENE AND PERIODONTAL CONDTION. Acta Odontol Scand. 1964 Feb;22:121-35. doi: 10.3109/00016356408993968. No abstract available. PMID 14158464
- [Background] Tian F, Mu H, Shi Y, Chen X, Zou X, Gao X, Wang X. Clinical evaluation of Giomer and self-etch adhesive compared with nanofilled resin composite and etch-and-rinse adhesive - Results at 8 years. Dent Mater. 2024 Jul;40(7):1088-1095. doi: 10.1016/j.dental.2024.05.013. Epub 2024 May 28. PMID 38806383
- [Background] Toz-Akalin T, Ozturk-Bozkurt F, Kusdemir M, Ozsoy A, Yuzbasioglu E, Ozcan M. Clinical Evaluation of Low-shrinkage Bioactive Material Giomer Versus Nanohybrid Resin Composite Restorations: A Two-year Prospective Controlled Clinical Trial. Oper Dent. 2023 Jan 1;48(1):10-20. doi: 10.2341/21-155-C. PMID 36508717
- [Background] Yadav G, Rehani U, Rana V. A Comparative Evaluation of Marginal Leakage of Different Restorative Materials in Deciduous Molars: An in vitro Study. Int J Clin Pediatr Dent. 2012 May;5(2):101-7. doi: 10.5005/jp-journals-10005-1145. Epub 2012 Aug 8. PMID 25206147